CLINICAL TRIAL: NCT01807195
Title: Acute Renal Injury Associated Contrast in Intensive Care Unit Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0922
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Acute Renal Injury
Keywords: contrast; Intensive care unit; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- the medical records of those in whom a contrast medium
  Interventions: Other: contrast medium usage

INTERVENTIONS:
Other: contrast medium usage

SUMMARY:
Generally, a contrast medium is used when performing a CT scan or radiographic tests such as angiography because it heightens image clarity and can increase diagnosis accuracy. Despite these advantages, contrast media can cause allergic reactions in the body or a decline in renal function. Therefore, they should be handled carefully and explained sufficiently to the patient. For intensive care patients, the use of contrast agents has been revealed as a major cause of acute renal damage, and many studies have investigated this complication by examining incidence rates and prevention strategies. Hypothesis: Among intensive care patients, the group in which a contrast medium was used will have a higher risk of renal function decline compared with the group in which a contrast medium was not used, and, hence, the use of contrast media becomes a cause of renal function deterioration. Categorizing patients with renal function decline according to the new RIFLE criteria can have an association with the prognosis of intensive care patients, such as hospitalization period and death rate, which can promote faster intervention.

ELIGIBILITY:
Inclusion Criteria:

* For the 5 years from January 2008 to December 2012, patients in whom a contrast medium was used in the intensive care unit were examined.

Exclusion Criteria:

* For the 5 years from January 2008 to December 2012, patients in whom a contrast medium was not used in the intensive care unit were examined.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RIFLE (Risk, Injury, Failure, Loss, and End-stage kidney disease) categorization and the existing classification method were used to compare their predictive value for acute renal damage related to contrast media.
Sampling Method: Non-Probability Sample
Enrollment: 886 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The incidence of acute renal damage associated with contrast media in intensive care patients | each time evaluation of contrast medium usage
  The occurrence of acute renal damage was examined, and these patients were compared with the group that did not develop acute renal damage to investigate whether the use of contrast agents acts as an independent variable. In addition, the RIFLE (Risk, Injury, Failure, Loss, and End-stage kidney disease) categorization and the existing classification method were used to compare their predictive value for acute renal damage related to contrast media.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim MH, Koh SO, Kim EJ, Cho JS, Na SW. Incidence and outcome of contrast-associated acute kidney injury assessed with Risk, Injury, Failure, Loss, and End-stage kidney disease (RIFLE) criteria in critically ill patients of medical and surgical intensive care units: a retrospective study. BMC Anesthesiol. 2015 Mar 3;15:23. doi: 10.1186/s12871-015-0008-x. eCollection 2015. PMID 25780349